CLINICAL TRIAL: NCT07278596
Title: Effect of High Intensity Focused Electromagnetic Therapy on Pain and Quality of Life in Patients With Lumbar Disc Prolapse: a Randomized Controlled Trial
Brief Title: High Intensity Focused Electromagnetic Therapy on Pain and Quality of Life in Patients With Lumbar Disc Prolapse
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Middle East University (Other)
Responsible Party: Principal Investigator, Saher Lotfy El Gayar, Assistant Professor of Physical Therapy, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Electromagnetic Therapy
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Back Pain Lower Back; Magnetic Therapy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity focused electromagnetic therapy group (Active Comparator): Participants in the study group will receive HIFEMT sessions using the HIFEMT device (Emsculpt Neo, BTL Industries, Boston, MA) twice weekly for 8 weeks.
  Interventions: Other: High intensity focused electromagnetic therapy (HIFEMT); Other: Stabilization exercise program
- Control group (Active Comparator): Stabilization Exercise Program:
  Both the study and control groups will receive lumbar stabilization exercise program three times weekly for 8 weeks.
  Interventions: Other: Stabilization exercise program

INTERVENTIONS:
Other: High intensity focused electromagnetic therapy (HIFEMT) — The patient will be positioned in a comfortable supine or seated position depending on the targeted lumbar area. The applicator will be placed over the lumbar spine, delivering focused electromagnetic pulses to stimulate deep core and paraspinal muscles. Each session will last 30 minutes, conducted three times per week over a period of 8 weeks. The intensity will be progressively adjusted according to patient tolerance, aiming to induce visible supramaximal muscle contractions without discomfort. HIFEMT is intended to promote muscle strengthening, pain modulation, and spinal stabilization.
  Arms: High intensity focused electromagnetic therapy group
Other: Stabilization exercise program — Participants will be guided through core-strengthening exercises aimed at improving trunk stability, posture, and neuromuscular control. The exercises will include pelvic tilts, bridging, and bird-dog exercises. All sessions will be conducted under supervision of a physiotherapist. Each session will last for approximately 30 minutes, three times weekly for 8 weeks.

SUMMARY:
Determine whether high intensity focused electromagnetic therapy has a significant effect on pain and quality of life in patients with lumbar disc prolapse.

DETAILED DESCRIPTION:
Lumbar disc prolapse is a common cause of lower back pain and radiculopathy, frequently affecting individuals in their productive years. It results from displacement of the intervertebral disc material beyond the disc space, leading to nerve root compression and significant pain, disability, and decreased quality of life. Persistent pain and reduced physical function can impair daily activities and may lead to psychological distress. Traditional conservative management, such as physical therapy and pharmacological interventions, may not always provide sufficient relief. High intensity focused electromagnetic therapy is a non-invasive modality that uses electromagnetic fields to stimulate deep muscle contractions. It has shown potential in enhancing muscle strength, modulating pain, and improving functional outcomes in musculoskeletal conditions. However, its role in managing lumbar disc prolapse has not been thoroughly investigated.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of lumbar disc prolapse by clinical and radiological evaluation.
* Ages between 30 and 60 years.
* A history of low back pain for at least three months.
* A body mass index less than 30 kg/m².

Exclusion Criteria:

* History of spinal surgery or recent traumatic spinal injury.
* Severe spinal canal stenosis or progressive neurological deficits.
* Known malignancy, infection, or inflammatory arthritis affecting the spine.
* Presence of implanted metal devices or pacemakers contraindicating electromagnetic therapy.
* Pregnancy or suspected pregnancy.
* Cognitive or psychological disorders that impair communication or ability to follow instructions

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-07 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Back pain | Baseline and after 8 weeks
  Using the Arabic Numerical Pain Rating Scale (NPRS) to evaluate the intensity of pain at baseline and post-intervention

SECONDARY OUTCOMES:
Quality of life assessment | Baseline and after 8 weeks
  Using the Short Form 12 Health Survey (SF-12) to evaluate both physical and mental health components of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sayed Saif, Study Director — National institute for Gerontology

IPD SHARING:
Plan to Share IPD: No